CLINICAL TRIAL: NCT03787940
Title: Optimizing Antituberculosis Therapy in Adults With Tuberculous Meningitis Based on N-Acetyltransferase Type 2 Genotyping
Brief Title: Optimizing Antituberculosis Therapy in Adults With Tuberculous Meningitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018ZX10302302-004
Record Dates: First submitted 2018-11-19; First posted 2018-12-27 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Tuberculous Meningitis
Keywords: N-Acetyltransferase Type 2 Genotype; treatment; Tuberculous Meningitis
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Isoniazid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard INH for Non-rapid acetylators (Active Comparator): Participant with slow or intermediate acetylators(one of N-Acetyltransferase Type 2 Genotype) administered with standard chemotherapy (3 months HRZE followed by 9 months HRE with standard dose isoniazid)
  Interventions: Drug: Isoniazid
- Standard INH for rapid acetylators (Active Comparator): Participant with rapid acetylators(one of N-Acetyltransferase Type 2 Genotype) administered with standard chemotherapy (3 months HRZE followed by 9 months HRE with standard dose isoniazid )
  Interventions: Drug: Isoniazid
- High dose INH for rapid acetylators (Experimental): Participant with rapid acetylators(one of N-Acetyltransferase Type 2 Genotype) administered with high dose isonized treatment (3 months HRZE followed by 9 months HRE with high dose isoniazid)
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: Isoniazid — standard dose isoniazid or high dose isoniazid for participants with rapid acetylators

SUMMARY:
The genetically polymorphic N-acetyltransferase type 2 (NAT2) is responsible for isoniazid metabolism, and rapid acetylators were associated with low concentrations of isoniazid based on previous studies. The investigators hypothesize that among rapid acetylators high dose isoniazid would result in lower rates of death and disability in patients with tuberculous meningitis than the rates with the standard regimen. The investigators recruited patients between the ages of 18 and 65 years with newly diagnosed TBM, then NAT2 genotype will be characterized by using High-Resolution Melting Kit (Zeesan Company, Xiamen). Participants with slow or intermediate acetylators will be administered with standard chemotherapy. For participants with rapid acetylators, patients were stratified at study entry according to the modified British Medical Research Council criteria (MRC grade), then randomly assigned in a 1:1 ratio to receive either standard or with high dose isoniazid treatment. All patients received antituberculosis treatment, which consisted of isoniazid (standard dose or high dose), rifampin, pyrazinamide, ethambutol for 3 months, followed by isoniazid, rifampin and ethambutol at the same doses for an additional 9 months. All patients received adjunctive treatment with dexamethasone for the first 6 to 8 weeks of treatment. 338 participants with rapid acetylators were randomly assigned to group B (standard treatment) and group C (high dose isoniazid), respectively. At the same time, 338 participants with slow or intermediate acetylators were recruited to group A (standard treatment). The primary outcome was death or severe disability 12 months after enrollment. Secondary outcome measures were coma-clearance time, fever-clearance time, and difference of laboratory examination (protein concentration, chloride, glucose and white cell counts) of cerebrospinal fluid.

DETAILED DESCRIPTION:
Tuberculous meningitis (TBM) is the most lethal form of tuberculosis, causing death or severe neurologic deficits in more than half of those affected in spite of antituberculosis chemotherapy. Among the first line drugs, isoniazid is the only bactericidal agent that easily crossed blood-brain barrier, achieving concentrations in cerebrospinal fluid (CSF) similar to those in serum. The genetically polymorphic N-acetyltransferase type 2 (NAT2) is responsible for isoniazid metabolism, and individuals can be classified as "rapid acetylators", "intermediate acetylators" or "slow acetylators" based on NAT2 genotyping. Rapid acetylators were associated with low concentrations of isoniazid based on previous studies. The investigators hypothesize that among rapid acetylators high dose isoniazid would result in lower rates of death and disability in patients with tuberculous meningitis than the rates with the standard regimen.

The investigators recruited patients between the ages of 18 and 65 years with newly diagnosed TBM. Patients could not enter the trial if they have been using any other second line antituberculosis drug; if they had received anti-tuberculosis therapy in the past 3 years；if they have positive CSF Gram or India ink stain; if they have received more than 14 days of anti-tuberculosis drugs for the current infection; if they were known or suspected hypersensitivity to or unacceptable side effects from any oral first line antituberculosis drug; if the plasma creatinine concentration was more than the upper limit of the normal range, if the plasma bilirubin concentration was more than 2 times the upper limit of the normal range, or if the plasma alanine aminotransferase level was more than three times the upper limit of the normal range; if they were known or suspected pregnancy; if they were known or suspected isoniazid and/or rifampin resistant; if they were lack of consent； if they were any participant for whom investigators judge this study is not appropriated.

Participants will be recruited from four sites in China, including Beijing Chest Hospital affiliated to Capital Medical University, Zunyi Medical College affiliated Hospital, Jiangxi Provincial Chest Hospital and Jiamusi Infectious Disease Hospital. All hospitals serve the local community and act as tertiary referral centers for patients with severe tuberculosis or infectious diseases in China.

Written informed consent to participate in the study was obtained from all patients. Then NAT2 genotype will be characterized by using High-Resolution Melting Kit (Zeesan Company, Xiamen). Participants with slow or intermediate acetylators will be administered with standard chemotherapy (3 months HRZE followed by 9 months HRE). For participants with rapid acetylators, patients were stratified at study entry according to the modified British Medical Research Council criteria (MRC grade), then randomly assigned in a 1:1 ratio to receive either standard or high dose isoniazid treatment.

All patients received antituberculosis treatment, which consisted of isoniazid (300 mg for standard treatment and 900 mg for high dose treatment), rifampin (450 mg for weight no more than 50 kg, 600 mg for weight more than 50 kg), pyrazinamide (1500 mg for weight no more than 50 kg, 1750 mg for weight more than 50 kg), ethambutol (750 mg for weight no more than 50 kg, 1000 mg for weight more than 50 kg) for 3 months, followed by isoniazid, rifampin and ethambutol at the same doses for an additional 9 months. All patients received adjunctive treatment with dexamethasone for the first 6 to 8 weeks of treatment, as recommend by British Infection Society.

338 participants with rapid acetylators will be randomly assigned to group B (standard treatment) and group C (high dose isoniazid), respectively. The calculation assumes an overall mortality and severe disability of 50% vs. 70 % in the two arms, a power of 80% and a two-sided significance level of 5%. Randomization ration is 1:1. At the same time, 338 participants with slow or intermediate acetylators were recruited to group A (standard treatment).

The primary outcome was death or severe disability 12 months after enrollment. Secondary outcome measures were coma-clearance time, fever-clearance time, and difference of CSF laboratory examination (protein concentration, chloride, glucose and white cell counts) of cerebrospinal fluid after 3 months treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age;
* Clinical diagnosis of TBM;
* Able and willing to provide informed consent to participate in the study.

Exclusion Criteria:

* Using any other second line antituberculosis drug;
* Received anti-tuberculosis therapy in the past 3 years；
* Positive CSF Gram or India ink stain;
* Received more than 14 days of anti-tuberculosis drugs for the current infection;
* Known or suspected hypersensitivity to or unacceptable side effects from any oral first line antituberculosis drug;
* Plasma creatinine concentration was more than the upper limit of the normal range, or the plasma bilirubin concentration was more than 2 times the upper limit of the normal range, or the plasma alanine aminotransferase level was more than three times the upper limit of the normal range;
* Known or suspected pregnancy;
* Known or suspected isoniazid and/or rifampin resistant;
* Lack of consent；
* Any participant for whom investigators judge this study is not appropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with death or severe disability | up to 12 months after enrollment
  Number of Participants with death or severe disability 12 months after enrollment

SECONDARY OUTCOMES:
days for coma-clearance time | through study completion,up to 1 year
  days for coma-clearance time through study completion
days for fever-clearance time | through study completion,up to 1 year
  days for fever-clearance time through study completion
difference of CSF protein concentration | 3 months after enrollment
  difference of CSF protein concentration (g/L)
difference of CSF glucose concentration | 3 months after enrollment
  difference of CSF glucose concentration (mmol/L)
difference of CSF white cell counts | 3 months after enrollment
  difference of CSF white cell counts (per milliliter)
difference of CSF chloride concentration | 3 months after enrollment
  difference of CSF chloride concentration (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Hongfei Duan, MD, Principal Investigator — Beijing Chest Hospital
Locations (4):
- China (4):
  - Beijing Chest Hospital affiliated to Capital Medical University, Beijing
  - Jiamusi Infectious Disease Hospital, Jiamusi
  - Jiangxi Provincial Chest Hospital, Nanchang
  - Zunyi Medical College affiliated Hospital, Zunyi

IPD SHARING:
Plan to Share IPD: Undecided